CLINICAL TRIAL: NCT06649513
Title: Long-term Ophthalmic Outcomes in Ex-premature Infants
Acronym: LTOO-XP
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Angela M. Arends-Tjiam, MD PhD, Pediatric Ophthalmologist, Erasmus Medical Center
Other Study IDs: 12793
Record Dates: First submitted 2024-09-20; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Retinopathy of Prematurity (ROP); Premature Birth
Keywords: Retinopathy of Prematurity; Preterm birth; Visual acuity; Visual outcomes; Long term outcomes
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preterm patients: Former patients who were born prematurely (GA < 37 weeks)
  Interventions: Diagnostic Test: eye drops (Tropicamid)

INTERVENTIONS:
Diagnostic Test: eye drops (Tropicamid) — Mydriatic + cycloplegic eye drops are given to measure refractive error and to image the full retina.

SUMMARY:
There is limited knowledge on ophthalmological outcomes in the adult population that was born prematurely. This study aims to evaluate the ophthalmic outcomes of ex-premature infants that have reached adolescence or adulthood.

DETAILED DESCRIPTION:
Every year, around 18.000 children in the Netherlands are born prematurely, which means that they were born before 37 weeks gestational age. The WHO defines three different categories of prematurity: moderate to late preterm (32-37 weeks), very preterm (<32-28 weeks), and extremely preterm (<28 weeks). Preterm birth is associated with numerous health problems, which can have both short-term and long-term consequences on the development of the child. A relatively rare complication of (very or extreme) preterm birth is lifelong visual impairment or blindness due to retinal detachment as a result of prematurity retinopathy (ROP). ROP is a vasoproliferative condition that affects the vessels in the retina. An inventory study shows that 305 children were diagnosed with ROP in the Netherlands in 2017. The majority of these children experienced spontaneous regression of the condition, but 13% of cases required treatment to prevent retinal detachment. In the long-term, ROP predisposes for ocular conditions such as visual field abnormalities, refractive error, strabismus, amblyopia, glaucoma and retinal detachment. However, research also indicates that prematurity, regardless of ROP diagnosis, can also be associated with adverse ophthalmological outcomes such as refractive error, strabismus, amblyopia and cerebral visual impairment (CVI). Although there are various publications on the ophthalmological outcomes of ROP and prematurity at school-age, less is known about these outcomes in the adult population. This study aims to investigate the anatomy and functionality of the eye in ex-premature infants who were born between 1991 and 2006. In addition, the differences in outcomes between ex-premature infants with and without ROP, and the differences in outcomes between treated and spontaneously regressed ROP, will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for ROP screening, and admitted to Erasmus MC between 1991 and 2007.

Exclusion Criteria:

* Subjects born after 2008,
* Subject has passed away before the start of the study
* Subject resides outside of the Netherlands
* Subject has a physical or mental disability that makes it impossible to participate in a routine eye exam, or has a disability that classifies the subject as an incapacitated adult.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature patients who were eligible for ROP screening, who were admitted to Erasmus MC between 1991 and 2007.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | The primary outcome measure will be assessed at one single visit to Erasmus MC. This one-off measurement will not be repeated, nor is there a specific time-frame for this measurement.
  Measured with ETDRS chart. Expressed in Logarithm of the Minimum Angle of Resolution (LogMAR)

SECONDARY OUTCOMES:
Biometric, refractive, fundus and Optical coherence tomography (OCT) data. | The secondary outcome measures will be assessed at one single visit to Erasmus MC. These one-off measurements will not be repeated, nor are there a specific time-frames for these measurements.
  * Refraction (spherical equivalent) in dioptre (D) measured with an automatic refractometer.
  * Optical biometry measurements (axial eye length in millimeters, lens thickness in millimeters, anterior chamber depth in millimeters) measured with an optical biometer.
  * Intra-ocular pressure (IOP) in millimeter in mercury (mmHg) measured with a non-contact or contact tonometer.
  * Visual field abnormalities measured with a Humphrey Field Analyzer (HFA), expressed as Visual Field Index (VFI), Mean Deviation (MD) and Pattern Standard Deviation (PSD) in decibels (dB).
  * Macula thickness in micrometers (µm) measured on Optical coherence tomography (OCT) images.
  * Any anatomical abnormalities of the retina and choroid seen on OCT of fundus images.
  * Presence of ophthalmological diagnoses such as amblyopia or strabismus.
  * Relevant (ophthalmological) medical history/ophthalmological diagnosis in the past.
  * Self-reported health, educational level, screen time and activity level (questionnaire).

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
We only plan to share anonymized and aggregated data.